CLINICAL TRIAL: NCT00634621
Title: A Post-authorization, Observational Study to Assess the Impact of Blue Light Cystoscopy After Administration of Hexaminolevulinate (Hexvix) in the Diagnosis and Treatment of Patients With Non-invasive Bladder Cancer.
Brief Title: Effectiveness of Hexaminolevulinate (Hexvix) in the Diagnosis and Treatment of Patients With Non-invasive Bladder Cancer
Status: Completed | Type: Observational
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: GEH-HEX-2007-01
Record Dates: First submitted 2008-02-26; First posted 2008-03-13 (Estimated); Results first posted 2014-08-25 (Estimated); Last update posted 2014-08-25 (Estimated); Status verified 2014-08

CONDITIONS: Bladder Cancer
Keywords: Bladder; Cancer; Cystoscopy; Hexaminolevulinate; Hexvix
MeSH Terms: conditions — Urinary Bladder Neoplasms; Neoplasms | interventions — 5-aminolevulinic acid hexyl ester

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Hexaminolevulinate (Hexvix) — Each patient enrolled into the study will be infused with 50 mL of a 2 mg/mL Hexvix solution in the bladder using a catheter. Subsequently, after fluid retention by the patient in the bladder for one hour, the bladder will be emptied.

SUMMARY:
The purpose of this study is to determine the effectiveness of hexaminolevulinate (Hexvix) in the diagnosis and treatment of patients with non-invasive bladder cancer and if it results in a change in patient management.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age.
* Patients of either sex.
* Patients with documented or highly suspected non-invasive bladder cancer.

Exclusion Criteria:

* Patients with hypersensitivity to the drug substance or any excipient of Hexvix.
* Patients with porphyry.
* Women of childbearing age.
* Patients at a high risk of suffering extensive bladder inflammation e.g. patients after intravesical BCG treatment, patients with moderate or severe leukocyturia or patients undergoing recent bladder surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with documented or suspected bladder cancer.
Sampling Method: Non-Probability Sample
Enrollment: 283 (Actual)
Dates: Start 2008-02; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Carlos Hernández, Principal Investigator — Gregorio Marañón Hospital, Madrid; Dr. Eduardo Solsona, Principal Investigator — Valencian Institute of Oncology, Valencia; Dr. Joan Palou, Principal Investigator — Fundación Puigvert, Barcelona
Locations (1):
- GE Healthcare, Madrid, Spain

RESULTS

PARTICIPANT FLOW:
Groups:
- Hexvix 2 mg/mL Infusion: Administrtation of 2 mg/mL Hexvix.
Period: Overall Study
Arm/Group | Hexvix 2 mg/mL Infusion
Started | 283
Completed | 283
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Hexvix: Use of the Hexvix drug.
Arm/Group | Hexvix
Number analyzed (Participants) | 283
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 110
  >=65 years | 173
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 243
Region of Enrollment [Number; unit: participants]
  Spain | 283

OUTCOME MEASURES:

1. Primary Outcome: Detecting the Rate of Bladder Cancer Lesions by White-Light Cystoscopy (WLC) and Blue-Light Cystoscopy (BLC) With Hexvix® in the Overall Study Population by Comparison With the Diagnostic Gold Standard, i.e. Histological Examination of Lesions Biopsy.
Description: Detecting the number of bladder cancer lesions by White-Light Cystoscopy (WLC) and Blue-Light Cystoscopy (BLC) with Hexvix®.
Time Frame: Day 0 (Post contrast administration)
Population: Number of True-positive lesions according to histology was 621 and broken out into various tumor stages. The Tumor stage distribution of true-positive bladder tumor lesions and their detection by White-light Cystoscopy (WLC) and/or Blue-light Cystoscopy (BLC).
Measure: Number; unit: Number of lesions
Groups:
- White-light and Blue-Light Cystoscopy Simultaneously: Hexvix administered using both White-light and Blue-Light Cystoscopy.
- White-light Cystoscopy Only: Hexvix administered using only White-light Cystoscopy.
- Blue-light Cystoscopy Only: Hexvix administered using only Blue-light Cystoscopy.
- Multiple Normalized Biopsy: Only Multiple Normalized Biopsy.
Arm/Group | White-light and Blue-Light Cystoscopy Simultaneously | White-light Cystoscopy Only | Blue-light Cystoscopy Only | Multiple Normalized Biopsy
Number analyzed (Participants) | 283 | 283 | 283 | 283
Number of lesions
  Tumor Stage-Carcinoma in situ | 41 | 1 | 31 | 30
  Tumor Stage-Ta | 236 | 2 | 64 | 1
  Tumor Stage- T1 | 127 | 0 | 9 | 2
  Tumor Stage- T2-T4 | 29 | 3 | 2 | 1
  Tumor could not be stage-Tx | 36 | 0 | 4 | 2
  TOTAL | 469 | 6 | 110 | 36

2. Secondary Outcome: Assess the Sensitivity of Standard White Light Cystoscopy (WLC) and Blue Light Cystoscopy (BLC) for Obtaining a Correct Diagnosis of Bladder Cancer at Individual Patient Level.
Description: The number of confirmed bladder cancer matches using cystoscopy compared to the diagnostic gold standard, i.e. histological examination of lesions biopsy.
Time Frame: Day 0 (Post contrast administration)
Population: The number of confirmed bladder cancer was 219 identified by the standard of truth methods using the White-light cystoscopy and blue-light cystoscopy technique.
Measure: Number (95% Confidence Interval); unit: Percentage of confirmed Lesions
Groups:
- Confirmed Bladder Cancer by Standard of Truth: Using the Hexvix drug with a cystoscopy technique of White-light cystoscopy and Blue-light cystoscopy.
Arm/Group | Confirmed Bladder Cancer by Standard of Truth
Number analyzed (Participants) | 283
Percentage of confirmed Lesions
  White-Light Cystoscopy-Sensitivity | 86.3 [81.7 to 90.9]
  Blue-Light Cystoscopy-Sensitivity | 90.9 [86.2 to 94.3]

ADVERSE EVENTS:
Arm/Group | Hexvix
Serious Adverse Events (participants affected / at risk) | 0/283
Other Adverse Events (participants affected / at risk) | 0/283

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No